CLINICAL TRIAL: NCT04061265
Title: Articaine Efficacy and Safety in Young Children Below Age of Four Years: An Equivalent Parallel Randomized Control Trial
Brief Title: Articaine Efficacy and Safety for Children Below Age of 4-years
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Ahmad Elheeny, Lecturer of Pediatri, Faculty of Dentistry, Minia University, Minia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 245
Record Dates: First submitted 2019-08-15; First posted 2019-08-19 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Behaviour Assessment; Pain
Keywords: Articaine, local anaesthesia, child, pain
MeSH Terms: conditions — Pain | interventions — Carticaine; Epinephrine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine 2% group (Active Comparator): lidocaine hydrochloride 2% and epinephrine 1:100000 (Lignospan® standard, 1.7ml, SEPTODONT Ltd)
  Interventions: Drug: lidocaine hydrochloride 2% and epinephrine 1:100000
- Articaine 4% (Experimental): articaine hydrochloride 4% and epinephrine 1:100000 (Septocaine® 1.7ml, SEPTODONT Ltd)
  Interventions: Drug: Articaine 4%/Epi 1:100000 Inj Cart 1.7Ml

INTERVENTIONS:
Drug: Articaine 4%/Epi 1:100000 Inj Cart 1.7Ml — Local anesthetic agent
  Arms: Articaine 4%
Drug: lidocaine hydrochloride 2% and epinephrine 1:100000 — Local anesthetic agent
  Arms: Lidocaine 2% group

SUMMARY:
Pain control is one of the significant behavior determinants in the dental office and shaping the future attitude toward dentistry, especially in children. One of widely used local anesthetic agents is articaine hydrochloride because of its superior potency, over traditionally used 2% lidocaine. Therefore, this study intends to get the benefits of articaine efficiency and apply it in children.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 36-47 months. ASA I, II. Mentally capable of communication. Having a mandibular primary molar tooth that required extraction or pulpotomy.

Exclusion Criteria:

* The presence of infection, which may compromise the efficiency of local anesthetic agent Significant behaviour problems Medical or mental unfitness

Ages: 37 Months to 47 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 184 (Actual)
Dates: Start 2019-08-25 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Pain assessment | During the procedures
  FLACC scale
Behavior | before and after the procedures
  Frankl behaviour scale

SECONDARY OUTCOMES:
postoperative complications | 24 hours after the procedures
  Asking parents/caregiver in the next 24 hours using Parents' postoperative pain measure (PPPM)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Elheeny, Principal Investigator — Cairo University
Locations (1):
- Ngwa Khattab, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No